CLINICAL TRIAL: NCT01389115
Title: Fatty Acids Lipidome and Oxidative Stress Markers as Indicators of Liver Transplant Outcome
Brief Title: Fatty Acids Lipidome and Oxidative Stress in Liver Transplantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Luigi Iuliano, M.D., University of Roma La Sapienza
Other Study IDs: Iul_LC
Record Dates: First submitted 2011-05-06; First posted 2011-07-07 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Liver Cirrhosis
Keywords: liver cirrhosis; oxidative stress; liver transplant
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples and liver biopsy specimens
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Liver Cirrhosis: Patient with liver cirrhosis undergoing liver transplant
- Liver donors: Subjects eligible for organ explant
- Healthy controls

SUMMARY:
The purpose of this study is to determine lipid metabolism in chronic liver disease in the attempt to find a useful biomarker of liver function and of prognostic value of graft function in those patients who undergo liver transplant. The present study enrolls subjects with liver cirrhosis (with different ethiology), including subjects eligible for a full-size liver transplantation, and healthy controls.

DETAILED DESCRIPTION:
Liver has a central role in fatty acids metabolism that is impaired in chronic liver diseases. Polyunsaturated fatty acids are reportedly reduced in liver cirrhosis, which is considered a condition of essential fatty acids deficiency. However, there is a paucity of data concerning the level of the multitude of circulating fatty acids in liver cirrhosis. Oxidative stress is involved in the pathogenesis of chronic liver disease and fibrosis. Increased oxidative stress with impaired antioxidant status at the systemic level has been described in different chronic liver diseases and negatively influences graft function after liver transplantation (Poli G. 2000, Loguercio C 2003). 7-Ketocholesterol and 7beta-hydroxycholesterol, prototype molecules of free radical-mediated cholesterol oxidation, are very important oxysterols currently accepted as in vivo reliable markers of oxidative stress. High oxysterols plasma levels are associated with an alteration of normal plasma fatty acid pattern in cystic fibrosis (Iuliano 2009). The Model for End-Stage Liver Disease (MELD) score is a common score used routinely to stage liver function in patients with liver cirrhosis (Al Sibae 2010). After ischemia-reperfusion injury at liver transplantation oxidative stress, hepatic endoplasmic reticulum (ER) stress and cholesterol metabolism are interrelated key processes to preserve graft regeneration and function. A blood sample is obtained in each subject to measure MELD score at the first visit and at liver transplantation. Further blood samples are collected at days seven and 30 post transplantation. Blood samples are also obtained from healthy subjects. Liver biopsy samples are obtained from liver transplant donors. Oxidative stress and fatty acids lipidomics are measured to evaluate the actual plasma concentration in liver cirrhosis patients to be compared with healthy controls. Oxidative stress and fatty acids are also analyzed as a function of disease status, and for its influence on transplant outcomes. Lipid metabolism gene and endoplasmic stress reticulum gene expression are evaluated in liver biopsy specimen to study the influence on graft function.

ELIGIBILITY:
Liver cirrhosis inclusion criteria:

* subjects with liver cirrhosis eligible for liver transplant, and one MELD score determination performed at least 3 months before liver transplantation

Liver cirrhosis exclusion criteria:

* liver transplant contraindication and re-transplantation
* current use of antioxidants and fatty acids supplements

Healthy controls are recruited recruited among the University personnel, after a review of their medical history.

Exclusion criteria for control participants included the use of drugs that affect fatty acids (systemic corticosteroids, isotretinoin, and ursodiol) and/or oxidative stress (antioxidants and hypolipemic drugs).

Ages: 15 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1. 150 cirrhotic patients, including Hepatocellular Carcinoma (HCC), Hepatitis C Virus (HCV) positive patients
  2. 80 healthy controls
  3. 100 liver donors
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2001-07; Primary Completion 2016-05 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Post operative graft function after liver transplantation | Change in graft function after 7 and 30 days after liver transplantation
  • Multiple lipid metabolism biomarkers (fatty acids, cholesterol and oxysterols) are evaluated in the plasma of liver cirrhosis patients before liver transplantation. A logistic regression model is used to evaluate which of these biomarkers is an independent predictor of graft function

SECONDARY OUTCOMES:
Early gene expression in the liver graft | 30 days
  Assessment of lipid metabolism-, oxidative stress-, and ER stress-gene expression in graft tissue liver tissue specimens of patients undergoing organ transplantation and their impact on graft function. Lipid metabolism and ER gene expression (genes: LDL-R, HMGCR, CD81, SREBP2, NPC1L1, XBP-1, XBP2, ATF6, GRP78, GRP94, LXR, INSIG1, INSIG2) in liver graft specimens at transplantation before and after ischemia-reperfusion injury; downregulated and upregulated genes are related to early graft function.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Corradini, M.D., Ph.D., Principal Investigator — University of Roma La Sapienza
Locations (3):
- Italy (3):
  - Department of Clinical Medicine Division of Gastroenterology, Sapienza University of Rome, Rome, RM
  - Liver Transplant Center Paride Stefanini, Sapienza University of Rome, Rome, RM
  - Laboratory of Vascular Medicine, Department of Medical Sciences and Biotechnology, Sapienza University of Rome, Latina

REFERENCES:
- [Background] Poli G. Pathogenesis of liver fibrosis: role of oxidative stress. Mol Aspects Med. 2000 Jun;21(3):49-98. doi: 10.1016/s0098-2997(00)00004-2. PMID 10978499
- [Background] Loguercio C, Federico A. Oxidative stress in viral and alcoholic hepatitis. Free Radic Biol Med. 2003 Jan 1;34(1):1-10. doi: 10.1016/s0891-5849(02)01167-x. PMID 12498974
- [Background] Iuliano L, Monticolo R, Straface G, Zullo S, Galli F, Boaz M, Quattrucci S. Association of cholesterol oxidation and abnormalities in fatty acid metabolism in cystic fibrosis. Am J Clin Nutr. 2009 Sep;90(3):477-84. doi: 10.3945/ajcn.2009.27757. Epub 2009 Jul 8. PMID 19587087
- [Background] Al Sibae MR, Cappell MS. Accuracy of MELD scores in predicting mortality in decompensated cirrhosis from variceal bleeding, hepatorenal syndrome, alcoholic hepatitis, or acute liver failure as well as mortality after non-transplant surgery or TIPS. Dig Dis Sci. 2011 Apr;56(4):977-87. doi: 10.1007/s10620-010-1390-3. Epub 2010 Sep 16. PMID 20844956
- [Result] Corradini SG, Micheletta F, Natoli S, Iappelli M, Di Angelantonio E, De Marco R, Elisei W, Siciliano M, Rossi M, Berloco P, Attili AF, Diczfalusy U, Iuliano L. High preoperative recipient plasma 7beta-hydroxycholesterol is associated with initial poor graft function after liver transplantation. Liver Transpl. 2005 Dec;11(12):1494-504. doi: 10.1002/lt.20524. PMID 16258953
- [Result] Iuliano L, Micheletta F, Natoli S, Ginanni Corradini S, Iappelli M, Elisei W, Giovannelli L, Violi F, Diczfalusy U. Measurement of oxysterols and alpha-tocopherol in plasma and tissue samples as indices of oxidant stress status. Anal Biochem. 2003 Jan 15;312(2):217-23. doi: 10.1016/s0003-2697(02)00467-0. PMID 12531208
- [Result] Corradini SG, Elisei W, De Marco R, Siciliano M, Iappelli M, Pugliese F, Ruberto F, Nudo F, Pretagostini R, Bussotti A, Mennini G, Eramo A, Liguori F, Merli M, Attili AF, Muda AO, Natalizi S, Berloco P, Rossi M. Preharvest donor hyperoxia predicts good early graft function and longer graft survival after liver transplantation. Liver Transpl. 2005 Feb;11(2):140-51. doi: 10.1002/lt.20339. PMID 15666381
- [Derived] Ginanni Corradini S, Zerbinati C, Maldarelli F, Palmaccio G, Parlati L, Bottaccioli AG, Molinaro A, Poli E, Boaz M, Serviddio G, Mennini G, Corsi A, Bianco P, Rossi M, Iuliano L. Plasma fatty acid lipidome is associated with cirrhosis prognosis and graft damage in liver transplantation. Am J Clin Nutr. 2014 Aug;100(2):600-8. doi: 10.3945/ajcn.113.074427. Epub 2014 Jun 25. PMID 24965302